CLINICAL TRIAL: NCT05817162
Title: Comparison of Temporomandibular Joint Arthrocentesis With Infiltration of PRP + Ropivacaine Versus PRP: Does It Reduce Postoperative Pain?
Brief Title: Temporomandibular Joint Arthrocentesis With Infiltration of PRP + Ropivacaine Versus PRP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Instituto Portugues da Face (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ROPIVACAINE_TMJ
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-03

CONDITIONS: Temporomandibular Joint Disorders
Keywords: temporomandibular disorders; temporomandibular joint arthrocentesis; ropivacaine; randomized clinical trial
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Ropivacaine; Arthrocentesis; Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: For this randomized clinical trial an appropriate number of sealed envelopes will be prepared: 15 for PRP and 15 for PRP + Ropivacaine. Patients with inclusion criteria will be seen in an orofacial pain session and assessed for pain using the VAS scale, by scoring the degree of pain between 0 (absence of pain) and 10 (maximum pain). Then the patients are proposed for TMJ arthrocentesis.
Who Masked: Investigator
Masking Description: The distribution of intervention is performed by attributing a code for each patient. Each code will have been previously distributed randomly between PRP + Ropicavaine and PRP only. The codes are kept closed singularly in an envelope. Before treatment, the nurse will ask the patient to choose an envelope. At this moment, the envelope is placed on a table, and the patient writes his name. Alone, the nurse opens the envelope and sees the code and the indication of PRP or PRP + Ropivacaine. Then, she will prepare, in her room, isolated from the whole team, one 3cc syringe with PRP or PRP + 1cc ropivacaine (7.5mg/ml), depending on the code. Once the code is attributed to the patient, she will deliver a tray with the prepared syringe for treatment. After finishing the arthrocentesis, the doctor injects the chosen treatment. Daily for one week, the patient answers a questionnaire, and at the end of the postoperative week, each patient will be blinded evaluated with a clinical examination.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group: PRP (Placebo Comparator): Temporomandibular joint arthrocentesis, Ringer lactate for washing, and 1ml PRP infiltration in each temporomandibular joint
  Interventions: Procedure: temporomandibular joint arthrocentesis; Drug: PRP injection; Drug: Ringer's Lactate solution
- PRP + Ropivacaine (Active Comparator): Temporomandibular joint arthrocentesis, Ringer lactate for washing, and 1ml PRP + ropivacaine infiltration in each temporomandibular joint
  Interventions: Drug: Ropivacaine injection; Procedure: temporomandibular joint arthrocentesis; Drug: PRP injection; Drug: Ringer's Lactate solution

INTERVENTIONS:
Drug: Ropivacaine injection — Ropivacaine is a local anesthetic that has been synthesized for use in infiltration anesthesia and to produce both peripheral and central block. Unlike one of its analogues, Bupivacaine, Ropivacaine anesthetize the sensory fibers without affecting the without affecting the motor ones. Ropivacaine comes as solution for injection.
  Arms: PRP + Ropivacaine
Procedure: temporomandibular joint arthrocentesis — Temporomandibular arthrocentesis is a minimally invasive surgical procedure, which aims to eliminate the inflammatory mediators from the inside of the TMJ.
Drug: PRP injection — Platelet-Rich Plasma (PRP) is an orthobiological adjuvant treatment. PRP has properties to restore intra-articular hyaluronic acid, increases glycosaminoglycan chondrocyte synthesis and balances joint angiogenesis. It is often used as a viscosupplement in TMJ arthrocentesis
Drug: Ringer's Lactate solution — Ringers lactate solution is used during arthrocentesis to wash out the joint inflammatory cells and to release the stuck disc phenomenon.

SUMMARY:
The infiltration of Platelet Rich Plasma (PRP) at the end of Temporomandibular Joint (TMJ) arthrocentesis is already an established procedure in the treatment of Temporomandibular Disorders (TMD). Arthrocentesis is a minimally invasive surgical procedure, which aims to eliminate the inflammatory mediators from the inside of the TMJ. PRP is an autologous concentrate of platelets and growth factors, derived from centrifugated blood. Several studies have described the benefits of PRP: it enhances wound healing because of the presence of cytokines and growth factors, and is also stimulates chondrocytes to biosynthesis of collagen. Ropivacaine is a local anesthetic that has been synthesized for use in infiltration anesthesia and to produce both peripheral and central block. Unlike one of its analogues, Bupivacaine, Ropivacaine anesthetize the sensory fibers without affecting the motor ones. The main goal of this investigation is to test the benefits of adding Ropivacaine to the infiltration of PRP in patients submitted to TMJ arthrocentesis.

DETAILED DESCRIPTION:
To investigate the potential reduction of pain in the postoperative week in patients submitted to temporomandibular joint double portal arthrocentesis with lavage and Platelet Rich Plasma (PRP) the authors designed a double-blind randomized clinical trial, comparing a treatment group with additional ropivacaine and a control group without ropivacaine.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between the ages of 18-99 years;
* For women of reproductive potential: use of highly effective contraception for at least 1 month prior to the first visit and agreement to use such a method during participation in the study;
* In the opinion of the investigator, the subject is capable of understanding and comprehending the study in question;
* The subject signs the written informed consent form and provides the necessary privacy clearance prior to the start of any study procedures;
* Patients with TMD with an indication for TMJ arthrocentesis: clinical and imaging diagnosis of unilateral or bilateral intra-articular disorder;
* Magnetic resonance imaging (MRI) assessing the intra-articular derangement;
* Radiological findings that most components of the joint were salvageable;
* Dimitroulis classification between 2 and 3.

Exclusion Criteria:

* Subject has had other previous minimally invasive or invasive treatment for TMD;
* Subject has any contraindication to the use of ropivacaine according to the Ropivacaine (Fresenius Kabi) bulletin;
* Subject has a history of allergy to any drug in the study;
* Subject taking analgesic medication prior to treatment for other conditions;
* The subject has an inability to interpret pain scales or to read and interpret the study's target questionnaire;
* Women who are pregnant or breastfeeding. For women of reproductive potential, use of highly effective contraception for at least 1 month prior to the first visit is required (Combined oral contraceptive pill, vaginal ring, male and female condom, intrauterine device, diaphragm, injectable hormonal contraceptive) and agreement to use such a method during study participation.
* Subjects under 18 and over 99 years old;
* Subjects diagnosed with the following conditions cannot participate in the study: cardiovascular disorders, peripheral vascular disease, arrhythmias, auriculoventricular conduction disorders, heart failure; hypotension, epileptic patients, patients with liver and kidney disease, patients with porphyria, patients with acidosis.
* Subjects with severe medical problems and mental illness.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
TMJ Pain | In the first week at a consultation after injection and TMJ arthrocentesis
  Change in TMJ pain in a 0-10 scale (where 0 is no pain and 10 is the maximum possible pain) assessed by the surgeon

SECONDARY OUTCOMES:
Postoperative pain | Daily 1 week after TMJ arthrocentesis and infiltration
  Change in TMJ pain / TMJ muscles pain: measured by the patient using a Visual Analogue scale (VAS), with a range from 0 to 10, with 0 being no pain and 10 having maximum unbearable pain. VAS score will be measured every day before TMJ arthrocentesis in the week after surgery.
General state pre vs post | Daily 1 week after TMJ arthrocentesis and infiltration
  Daily questionnaire based (OHIP 10) furnished by surgeon to fill at home: the patient has to fill it every day for 1 week. (0-much better, 1-litte better, 2-no changes, 3-litter worse, 4-much worse)
Functional limitation chewing foods | Daily 1 week after TMJ arthrocentesis and infiltration
  Daily questionnaire based (OHIP 10) furnished by surgeon to fill at home: the patient has to fill it every day for 1 week (0-never, 1-hardly never, 2-occasionally, 3-fairy often, 4-very often)
Difficulty closing and mouth opening | Daily 1 week after TMJ arthrocentesis and infiltration
  Daily questionnaire based (OHIP 10) furnished by surgeon to fill at home: the patient has to fill it every day for 1 week (0-never, 1-hardly never, 2-occasionally, 3-fairy often, 4-very often)
TMJ pain, muscular pain, ear pain | Daily 1 week after TMJ arthrocentesis and infiltration
  Daily questionnaire based (OHIP 10) furnished by surgeon to fill at home: the patient has to fill it every day for 1 week (0-never, 1-hardly never, 2-occasionally, 3-fairy often, 4-very often)
Interrupt meals | Daily 1 week after TMJ arthrocentesis and infiltration
  Daily questionnaire based (OHIP 10) furnished by surgeon to fill at home: the patient has to fill it every day for 1 week (0-never, 1-hardly never, 2-occasionally, 3-fairy often, 4-very often)
Sleep been interrupted | Daily 1 week after TMJ arthrocentesis and infiltration
  Daily questionnaire based (OHIP 10) furnished by surgeon to fill at home: the patient has to fill it every day for 1 week (0-never, 1-hardly never, 2-occasionally, 3-fairy often, 4-very often)
Difficult doing usual jobs | Daily 1 week after TMJ arthrocentesis and infiltration
  Daily questionnaire based (OHIP 10) furnished by surgeon to fill at home: the patient has to fill it every day for 1 week (0-never, 1-hardly never, 2-occasionally, 3-fairy often, 4-very often)
Unable to work full capacity | Daily 1 week after TMJ arthrocentesis and infiltration
  Daily questionnaire based (OHIP 10) furnished by surgeon to fill at home: the patient has to fill it every day for 1 week (0-never, 1-hardly never, 2-occasionally, 3-fairy often, 4-very often)
Difficult to relax | Daily 1 week after TMJ arthrocentesis and infiltration
  Daily questionnaire based (OHIP 10) furnished by surgeon to fill at home: the patient has to fill it every day for 1 week (0-never, 1-hardly never, 2-occasionally, 3-fairy often, 4-very often)
Need of medication after intervention | Daily 1 week after TMJ arthrocentesis and infiltration
  Indication of the number of SOS analgesic pills taken each day
TMJ pain assessed by the physiotherapist | 1 week after injection and TMJ arthrocentesis in a physiotherapy consultation
  Pain in left and right TMJ evaluated by the physiotherapist in a 0-10 scale (where 0 is no pain and 10 is the maximum possible pain)
TMJ pain during lateral deviation assessed by the physiotherapist | 1 week after injection and TMJ arthrocentesis in a physiotherapy consultation
  Pain in left and right TMJ during lateral deviation evaluated by the physiotherapist in a 0-10 scale (where 0 is no pain and 10 is the maximum possible pain)
TMJ pain during protrusion assessed by the physiotherapist | 1 week after injection and TMJ arthrocentesis in a physiotherapy consultation
  TMJ pain during protrusion evaluated by the physiotherapist in a 0-10 scale (where 0 is no pain and 10 is the maximum possible pain)
Myalgia degree assessed by the physiotherapist | 1 week after injection and TMJ arthrocentesis in a physiotherapy consultation
  Myalgia degree in right and left masseter and temporalis muscles evaluated by the physiotherapist in a 0-3 scale
Physiotherapist's perception of comfort during the consultation | 1 week after injection and TMJ arthrocentesis in a physiotherapy consultation
  For the therapist: in a 0 to 10 scale evaluate your perception of patients comfort during the physical therapy question

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Português da Face, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No
Due to data protection policy it is not possible to share this data with other researchers.

REFERENCES:
- [Background] Derwich M, Mitus-Kenig M, Pawlowska E. Mechanisms of Action and Efficacy of Hyaluronic Acid, Corticosteroids and Platelet-Rich Plasma in the Treatment of Temporomandibular Joint Osteoarthritis-A Systematic Review. Int J Mol Sci. 2021 Jul 9;22(14):7405. doi: 10.3390/ijms22147405. PMID 34299024
- [Background] Keyser C, Bhashyam A, Abdurrob A, Smith JT, Bluman E, Chiodo C. Excess Opioid Disposal Following Orthopaedic Surgery: A Randomized Clinical Trial. Foot Ankle Spec. 2022 Dec;15(6):545-550. doi: 10.1177/1938640020980921. Epub 2020 Dec 27. PMID 33356547
- [Background] Rao TN, Goswami D, Roychoudhury A, Bhutia O, Baidya DK, Trikha A. Efficacy of Local Anesthetic Wound Infiltration in Temporomandibular Joint Ankylosis Surgery for Control of Postoperative Pain: A Prospective, Randomized Controlled, and Double-Blinded Trial. J Oral Maxillofac Surg. 2021 Mar;79(3):559.e1-559.e11. doi: 10.1016/j.joms.2020.10.034. Epub 2020 Oct 29. PMID 33232658

DOCUMENTS (1):
  • Informed Consent Form (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT05817162/ICF_000.pdf